CLINICAL TRIAL: NCT04494295
Title: The MIRROR Registry: Minimally Invasive IntRaceRebral HemORrhage Evacuation
Acronym: MIRROR
Status: Recruiting | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Oculus Imaging LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: C-MIRROR-001
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Supratentorial Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- AURORA: Aurora® Surgiscope used for MIS evacuation of supratentorial hematoma
  Interventions: Device: Aurora Surgiscope System

INTERVENTIONS:
Device: Aurora Surgiscope System — MIS evacuation of hematoma using the Aurora Surgiscope System

SUMMARY:
This registry will study the use of the Aurora® Surgiscope to provide surgical access and visualization in minimally invasive removal of hematoma in the brain. Many methods of hematoma removal are available and will be based on surgeon preference. The impact of patient selection and time to surgery from last known well time will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Subject Age is > 18
* Subject with a Head CT that demonstrates an acute, spontaneous, primary, supratentorial ICH of volume > 20 mL, assessed via standard of care techniques
* Subject Surgery can be initiated within 24 hours of the last known well time or, in patients with wake-up onset, within 24 hours of the time the patient awoke with symptoms.
* Subject has a NIHSS score > 5
* Subject has a baseline Modified Rankin Scale (mRS) Score ≤ 2
* Subject with a CT Angiography demonstrating no vascular malformation

Exclusion Criteria:

* Subject has an underlying vascular lesion defined as causative source of ICH
* Subject has a profound neurological deficit defined as fixed/dilated pupils or bilateral extensor motor posturing
* Subject has an Infratentorial or brainstem ICH
* Subject has a known life expectancy < 6 months
* Subject has an uncorrectable coagulopathy
* Subject has a mechanical heart valve
* Subject is pregnant
* Subject participates in another concurrent interventional clinical trial
* Subject who is unable to meet study follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: general population with an acute, spontaneous, primary, supratentorial ICH
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2028-10-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
Rate of Surgical Success | During surgical procedure to evacuate supratentorial intracerebral hemorrhage
  Rate of surgical success defined as reduction to < 15 cc total volume of the supratentorial intracerebral hemorrhage on immediate Post-op CT Scan

CONTACTS AND LOCATIONS:
Overall Officials: Sigmund Kulessa, Study Director — Integra LifeSciences Corporation; Christopher Kellner, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (20):
- United States (20):
  - Providence Health, Burbank, California
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - MedStar Health Research Institute, Baltimore, Maryland
  - Corewell Health, Grand Rapids, Michigan
  - University of Missouri, Columbia, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - JFK university, Edison, New Jersey
  - University at Buffalo, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Prisma Health - Upstate, Greenville, South Carolina
  - UT Health, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington - Harborview, Seattle, Washington